CLINICAL TRIAL: NCT07227402
Title: A Phase 3, Randomized, Open-label Study of Belzutifan + Zanzalintinib Versus Cabozantinib in Participants With Advanced RCC Who Experienced Disease Recurrence During or After Prior Adjuvant Anti-PD-1/L1 Therapy (LITESPARK-033)
Brief Title: A Clinical Study of Belzutifan and Zanzalintinib in People With Recurrent Kidney Cancer Following Adjuvant Therapy (MK-6482-033)
Acronym: LITESPARK-033
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-033; U1111-1311-6892 (Registry Identifier: UTN); 2024-517136-21 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Carcinoma; Renal cell; Belzutifan; Zanzalintinib
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma | interventions — belzutifan; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan plus Zanzalintinib (Experimental): Participants will receive belzutifan orally once daily (QD) PLUS zanzalintinib orally QD until one of the reasons for discontinuation of study intervention are met.
  Interventions: Drug: Belzutifan; Drug: Zanzalintinib
- Cabozantinib (Active Comparator): Participants will receive cabozantinib orally QD until one of the reasons for discontinuation of study intervention are met.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Belzutifan — Administered orally QD
  Other Names: MK-6482; PT2977; WELIREG™
  Arms: Belzutifan plus Zanzalintinib
Drug: Zanzalintinib — Administered orally QD
  Other Names: XL092
  Arms: Belzutifan plus Zanzalintinib
Drug: Cabozantinib — Administered orally QD
  Arms: Cabozantinib

SUMMARY:
Researchers are looking for more ways to treat advanced renal cell carcinoma (RCC) that is recurrent. Researchers want to learn if recurrent advanced renal cell carcinoma (RCC) responds (gets smaller or goes away) after treatment with belzutifan (MK-6482) and zanzalintinib compared to cabozantinib.

The goal of this study is to learn if:

People who take belzutifan and zanzalintinib live longer overall and without the cancer getting worse than people who take cabozantinib.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a histologically confirmed diagnosis of unresectable, advanced renal cell cancer (RCC) with clear cell component (with or without sarcomatoid features) i.e., Stage IV renal cell cancer per American Joint Committee on Cancer (AJCC) (8th Edition)
* Has measurable disease per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
* Has disease recurrence during adjuvant anti-programmed cell death 1/programmed cell death ligand 1 (PD-1/L1) therapy or recurrence ≤24 months following the last dose of adjuvant anti-PD-1/L1 therapy
* Has received no other prior systemic therapy for their RCC except for their adjuvant anti-PD-1/L1 therapy

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, new-onset angina, pulmonary embolism, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Had deep vein thrombosis within 3 months before randomization unless stable, asymptomatic, and treated with therapeutic anticoagulation for at least 4 weeks before randomization
* Has a left ventricular ejection fraction ≤50% or below the institutional (or local laboratory) normal range as determined by multigated acquisition or echocardiogram
* Has had major surgery within 8 weeks before randomization or has not adequately recovered from major surgery or has ongoing surgical complications
* Has current pneumonitis/interstitial lung disease
* Has symptomatic pleural effusion (for example cough, dyspnea, pleuritic chest pain), ascites, or pericardial fluid requiring drainage within 4 weeks prior to randomization
* Has a gastrointestinal disorder including those associated with a high risk of perforation or fistula formation
* Has a serious active nonhealing wound/ulcer/bone fracture
* Has a requirement for hemodialysis or peritoneal dialysis
* Has history of human immunodeficiency virus infection
* Has hepatitis B or hepatitis C virus
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2032-02-27 (Estimated); Study Completion 2032-02-27 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 73 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PD will be assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Overall Survival (OS) | Up to approximately 73 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 73 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Duration of Response (DOR) | Up to approximately 73 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by Blinded Independent Central Review (BICR) will be presented.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 73 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Number of Participants Who Discontinue Study Treatment due to an AE | Up to approximately 73 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue the study treatment due to an AE will be reported.
Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC QLQ-C30) Global Health/Health-Related Quality of Life (HRQoL) Items 29 and 30 Combined Score | Up to approximately 25 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent), then summed. Summed raw scores are standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome.
Change From Baseline in EORTC QLC-C30 Physical Functioning Items 1-5 Score | Up to approximately 25 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome.
Change From Baseline in EORTC QLQ-C30 Role Functioning Items 6-7 Score | Up to approximately 25 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Summed raw scores are standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better level of functioning.
Change From Baseline in Functional Assessment of Cancer Therapy-Kidney Symptom Index-Disease-related Symptoms (FKSI-DRS) Items 1-9 Score | Up to approximately 25 months
  The FKSI-DRS index consists of a 9-item questionnaire that assesses the extent of participant symptoms from kidney cancer. Responses are scored on a 5-point scale (0=Not at all to 4=Very much) and summed to generate an index symptom score. These scores can range from 0 to 36, with a higher score indicating more favorable kidney cancer symptom status.
Time From Baseline to First Deterioration in EORTC-QLC-C30 Global Health/HRQoL Score | Up to approximately 25 months
  Time to True Deterioration (TTD) is defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in Items 29 and 30 scale scores. A longer TTD indicates a better outcome. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time From Baseline to First Deterioration in EORTC-QLC-C30 Physical Functioning Score | Up to approximately 25 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point deterioration (decrease) from baseline in physical functioning score (EORTC QLQ-C30 Items 1-5). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in physical functioning score will be presented. A longer TTD indicates a better outcome.
Time From Baseline to First Deterioration in EORTC-QLC-C30 Role Functioning Score | Up to approximately 25 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in role functioning (EORTC QLQ-C30 Items 6 and 7) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in role functioning score, will be presented. A longer TTD indicates a better outcome.
Time From Baseline to First Deterioration in FKSI-DRS Score | Up to approximately 25 months
  TTD is defined as time from the first dose of study treatment to the date of deterioration of FKSI-DRS Score. Each item is scored on a 5-point scale (0=not at all to 4=very much). FKSI-DRS total score ranged from 0 (most severe symptoms) to 36 (no symptoms) with a higher score indicating a better outcome. Deterioration is defined as a 3-point decrease (i.e. lower score) in symptom score and the time to true deterioration is the time to first onset of 3 or more decreases from baseline with confirmation under right-censoring rule (the last observation). A longer TTD indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (75):
- Argentina (5):
  - Asociación de Beneficencia Hospital Sirio Libanés ( Site 0205), Caba, Buenos Aires
  - Instituto Alexander Fleming ( Site 0202), CABA, Buenos Aires
  - Sanatorio Parque ( Site 0201), Rosario, Santa Fe Province
  - Instituto de Oncología de Rosario ( Site 0209), Rosario, Santa Fe Province
  - Hospital Privado Universitario de Córdoba ( Site 0207), Córdoba
- Macquarie University-MQ Health Clinical Trials Unit ( Site 2100), Sydney, New South Wales, Australia
- Ordensklinikum Linz GmbH Elisabethinen-Urologie ( Site 0600), Linz, Upper Austria, Austria
- Belgium (4):
  - Cliniques Universitaires Saint-Luc ( Site 0703), Brussels, Bruxelles-Capitale, Region de
  - Ziekenhuis Oost-Limburg, Campus St.-Jan ( Site 0701), Genk, Limburg
  - UZ Gent ( Site 0702), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0700), Leuven, Vlaams-Brabant
- Czechia (6):
  - Masarykuv onkologicky ustav ( Site 0903), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava ( Site 0904), Ostrava, Ostrava Mesto
  - Nemocnice České Budějovice ( Site 0905), České Budějovice
  - Fakultni nemocnice Hradec Kralove ( Site 0902), Hradec Králové
  - Fakultni nemocnice Olomouc ( Site 0901), Olomouc
  - Fakultni nemocnice v Motole ( Site 0900), Prague
- Denmark (2):
  - Herlev Hospital ( Site 1002), Herlev, Capital Region
  - Odense Universitetshospital ( Site 1000), Odense, Region Syddanmark
- France (9):
  - CHU de Bordeaux Hop St ANDRE ( Site 1115), Bordeaux, Gironde
  - Hôpital Foch ( Site 1118), Suresnes, Hauts-de-Seine
  - Centre de Cancérologie du Grand Montpellier ( Site 1112), Montpellier, Herault
  - CHU GRENOBLE ALPES ( Site 1101), La Tronche, Isere
  - Centre d'Oncologie de Gentilly ( Site 1117), Nancy, Lorraine
  - Centre Hospitalier Universitaire d'Angers-Urology ( Site 1104), Angers, Pays de la Loire Region
  - Centre Hospitalier de la Côte Basque ( Site 1113), Bayonne, Pyrenees-Atlantiques
  - HENRI MONDOR HOSPITAL ( Site 1116), Créteil, Val-de-Marne
  - CHD Vendee ( Site 1103), La Roche-sur-Yon, Vendee
- Germany (7):
  - Klinikum Stuttgart - Katharinenhospital ( Site 1201), Stuttgart, Baden-Wurttemberg
  - Universitätsmedizin Göttingen - Georg-August-Universität ( Site 1211), Göttingen, Lower Saxony
  - Helios Kliniken Schwerin GmbH ( Site 1206), Schwerin, Mecklenburg-Vorpommern
  - Universitaetsklinikum Muenster ( Site 1202), Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden ( Site 1213), Dresden, Saxony
  - HELIOS Klinikum Erfurt ( Site 1208), Erfurt, Thuringia
  - Universitätsklinikum Jena ( Site 1204), Jena, Thuringia
- Greece (2):
  - Alexandra General Hospital of Athens ( Site 1300), Athens, Attica
  - Metropolitan Hospital ( Site 1302), Athens, Attica
- Hong Kong (2):
  - Prince of Wales Hospital ( Site 2200), Hong Kong
  - Queen Mary Hospital ( Site 2201), Hong Kong
- Italy (7):
  - Istituto Nazionale Tumori Regina Elena ( Site 1611), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1600), Milan, Milano
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1601), Rome, Roma
  - Azienda Ospedaliera Universitaria Careggi ( Site 1608), Florence, Tuscany
  - Casa di Cura Dott. Pederzoli - UO Oncologia ( Site 1610), Peschiera del Garda, Veneto
  - Azienda USL 8 di Arezzo ( Site 1605), Arezzo
  - Ospedale San Martino ( Site 1606), Genova
- Mexico (5):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0503), Guadalajara, Jalisco
  - I CAN ONCOLOGY CENTER S.A. DE C.V. ( Site 0507), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0502), Oaxaca City, Oaxaca
  - Higiea Oncologia ( Site 0504), Mexico City
  - Clinica Integral Internacional de Oncología ( Site 0506), Puebla City
- Poland (4):
  - Pratia MCM Krakow ( Site 1713), Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 1703), Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1702), Siedlce, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1710), Przemyśl, Podkarpackie Voivodeship
- National Cancer Centre Singapore ( Site 2401), Singapore, Central Singapore, Singapore
- South Korea (5):
  - Chonnam National University Hwasun Hospital ( Site 2505), Hwasun-gun, Jeonranamdo
  - Seoul National University Bundang Hospital ( Site 2504), Seongnam, Kyonggi-do
  - Chungnam National University Hospital ( Site 2506), Taejŏn, Taejon-Kwangyokshi
  - Severance Hospital, Yonsei University Health System ( Site 2503), Seoul
  - Samsung Medical Center ( Site 2502), Seoul
- Spain (10):
  - Hospital Universitario Marqués de Valdecilla ( Site 1807), Santander, Cantabria
  - Institut Català d'Oncologia (ICO) - Girona ( Site 1806), Girona, Gerona
  - Hospital Universitario Ramón y Cajal ( Site 1801), Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología ( Site 1808), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron ( Site 1804), Barcelona
  - Hospital Clinic de Barcelona ( Site 1810), Barcelona
  - Hospital Universitario Reina Sofia ( Site 1809), Córdoba
  - Hospital Clinico San Carlos ( Site 1802), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 1803), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1800), Madrid
- Taiwan (4):
  - China Medical University Hospital ( Site 2603), Taichung
  - Taichung Veterans General Hospital ( Site 2602), Taichung
  - Taipei Veterans General Hospital ( Site 2600), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 2604), Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/